CLINICAL TRIAL: NCT05542875
Title: Effects of Thrust Versus Non-Thrust Thoracic Manipulation on Mechanical Neck Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/15
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Thrust Manipulation) (Experimental): Participants will be randomly allocated to Group A which will recieve Thrust manipulation treatment in addition to standard treatment protocol. Prone thoracic extension manipulation technique will be applied from T2 - T6 to participants for 4 sessions on alternate days
  Interventions: Procedure: Thrust Manipulation; Procedure: Standard Treatment
- Group B (Non-Thrust Manipulation) (Experimental): Participants will be randomly allocated to group B which, in addition to standard treatment protocol, will recieve Maitland grade III or IV manipulation from T1 to T6. Posterior to anterior glide over spinous process will be maintained for 30 seconds. Participants will recieve 4 sessions on alternate days
  Interventions: Procedure: Non-Thrust manipulation; Procedure: Standard Treatment

INTERVENTIONS:
Procedure: Thrust Manipulation — Prone thoracic extension manipulation technique will be applied from T2 - T6 to participants of Group A (Experimental group). Intervention will be applied on alternate days with a total of 4 treatment sessions
  Arms: Group A (Thrust Manipulation)
Procedure: Non-Thrust manipulation — Maitland grade III or IV thoracic 0manipulation will be given to participants of Control group from T1 to T6. Posterior to anterior glide over spinous process will be maintained for 30 seconds. Intervention will be applied on alternate days with a total of 4 treatment sessions
  Arms: Group B (Non-Thrust Manipulation)
Procedure: Standard Treatment — Standard treatment protocol includes moist heat, TENS and Post isometric relaxation technique. Standard treatment will be given to both groups on every session. Standard treatment consists of:
  Superficial Moist Heat (Device): Superficial moist heat will me applied for 10 minutes on Upper Trapezius TENS (Device): TENS will be applied for 10 minutes at 80-100Hz, the electrodes will be placed at upper trapezius.
  Post-isometric Relaxation (procedure/surgery): 5-10 repetions of Post Isometric relaxation technique will be applied on various muscle groups which include Upper trapezius, levator scapulae, sternocleidomastoid and scalenes.

SUMMARY:
Neck pain ranks as the 4th leading cause of disability, with high prevalence of mechanical neck pain in young population. As high as 30% of %. Individuals suffering from neck often report difficulty in performance of daily life, absence from work and decreased productivity. Several manual therapy treatment approaches are used for mechanical neck pain. The focus of this study is to compare the effectiveness of thrust and non-thrust thoracic manipulation for the treatment of mechanical neck pain in young population

DETAILED DESCRIPTION:
craniovertebral angle, cervical range of motion and pain will be noted for each participant.

ELIGIBILITY:
Inclusion Criteria

* Both genders
* Age: 18-24 years
* Symptoms <30 days
* FABQPA score <12
* Increased upper thoracic spine kyphosis (visual estimate)
* CVA < 48 Degrees

Exclusion Criteria

* Symptoms distal to shoulder
* Aggravation of symptoms with looking up
* Radiating lower back pain
* Neurological deficit
* Previous surgery
* Spondylolisthesis
* Spinal stenosis
* Inflammatory disease
* Vertebrobasilar artery insufficiency
* Pregnancy

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral Angle | 8 days
  Craniovertebral Angle wll be measured using Goniometer. CVA >48 is considered normal, CVA <48 is considered as Forward head posture. Immovable arm of the goniometer will be placed at the C7 spinous process and the movable arm at the tragus of the ear making an angle between the two lines, normal of which is 49.9 and angle less than that is considered as abnormal. Data will be collected directly from participants using Gomiometer before initiation of treatment and after 4th session.

SECONDARY OUTCOMES:
Cervical Range of Motion | 8 days
  Cervical Range of motion will be measured using bubble inclinometer. Measurement will be taken before the initiation of treatment and after 4Th treatment session. Increase in Cervical ROM will be considered a positive outcome.
Pain intensity | 8 days
  Pain will be assessed using Numeric pain rating scale which comprises of 11 points where point (0) signifies no pain and point (10) signifies worst imaginable pain. Measurement will be taken before the initiation of treatment and after 4Th treatment session. Low score for the NPRS will be considered a positive outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan